CLINICAL TRIAL: NCT02078609
Title: A Phase I, Multicenter, Open-label Study of Oral LGH447 in Patients With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Brief Title: A Safety and Efficacy Study of LGH447 in Patients With Acute Myeloid Leukemia (AML) or High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLGH447X2102; 2013-003756-20 (EudraCT Number)
Record Dates: First submitted 2014-01-31; First posted 2014-03-05 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-01

CONDITIONS: AML and High Risk MDS
Keywords: AML,; MDS,; PIM,; LGH447,; acute myelod leukemia,; myelodysplastic syndrome,; midostaurin,; PKC412
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — LGH-447; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LGH447 monotherapy arm (Experimental): LGH447 monotherapy in patients with AML or MDS
  Interventions: Drug: LGH447
- LGH447 + midostaurin combination arm (Experimental): LGH447 + midostaurin in patients with AML
  Interventions: Drug: LGH447 + midostaurin

INTERVENTIONS:
Drug: LGH447 — LGH447 in patients with AML or MDS
  Arms: LGH447 monotherapy arm
Drug: LGH447 + midostaurin — LGH447 + midostaurin in patients with AML
  Arms: LGH447 + midostaurin combination arm

SUMMARY:
This study will assess the safety and preliminary efficacy of escalating doses of LGH447 monotherapy in AML and MDS and LGH447 in combination with midostaurin in AML.

ELIGIBILITY:
Inclusion Criteria

-Male or female patients ≥18 years of age who present with one of the following:

LGH447 monotherapy arm

* Refractory/Relapsed AML following no more than 2 prior therapies, or in previously untreated AML patients who are not candidates for standard therapy.
* High and very high risk MDS according to the revised International Prognostic Scoring System (rIPSS) who have failed prior therapies, such as azacitidine and decitabine
* Patients with rIPSS score of > 4.5

LGH447 and midostaurin combination arm

* Refractory/Relapsed AML following no more than 2 prior therapies, or in previously untreated AML patients who are not candidates for standard therapy. AML patients may have either FLT3 wild type or FLT3-ITD/TKD mutant disease, and FLT3 mutation status needs to be defined at study entry.

  * For AML patients, peripheral blast counts < 50,000 blasts/mm3
  * For MDS patients;
* Platelet count > 25,000/mm3
* Neutrophils > 500/mm3
* Blood transfusions are allowed to maintain clinically adequate hemoglobin and hematocrit levels

  * Patients with active central nervous system (CNS) disease are eligible to participate and may be treated concurrently with intrathecal (or intra Ommaya) chemotherapy
  * Patients who are maintained on prophylactic antibiotics are eligible to participate as long as agents comply with the list of approved concomitant medications
  * Performance status ≤ 2
  * Meet other lab criteria

Exclusion Criteria

* Systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any experimental therapy within 7 days or 5 half-lives, whichever is longer, before the first dose of LGH447 monotherapy or LGH447 in combination with midostaurin
* Radiotherapy with a wide field of radiation within 28 days or radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of LGH447 monotherapy or LGH447 in combination with midostaurin
* Patients who received CNS irradiation for meningeal leukemia, except if radiotherapy occurred > 3 months previously
* Major surgery within 4 weeks before the first dose of LGH447 monotherapy or LGH447 in combination with midostaurin
* Ongoing therapy with corticosteroids greater than 10 mg of prednisone or its equivalent per day. Inhaled and topical steroids are permitted
* Patients who are currently receiving hydroxyurea to control peripheral blood leukemic blasts and cannot be discontinued for at least 48 hours prior to obtaining PD biomarkers at screening/baseline and during the study
* Patients who are currently receiving treatment with prohibited medication and that cannot be discontinued at least one week prior to the start of treatment with LGH447 monotherapy or LGH447 in combination with midostaurin
* Active infection requiring systemic therapy or other severe infection, including pneumonia, within 2 weeks before the first dose of LGH447 monotherapy or LGH447 in combination with midostaurin
* Known human immunodeficiency virus (HIV) positive
* Corrected QT interval (QTc) of > 450 milliseconds (ms) in males and > 470 milliseconds (ms) in females on baseline electrocardiogram (ECG) (using corrected QT interval using Fridericia [QTcF] or local standards).
* Uncontrolled cardiovascular condition, including ongoing cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) of LGH447 monotherapy arm in patients with AML or MDS and of LGH447 + midostaurin in patients with AML | 28 days post study treatment
  Frequency and characteristics of dose limiting toxicities

SECONDARY OUTCOMES:
Number of participants with the type, frequency, and severity of adverse events (AEs) as a measure of safety and tolerability of the LGH447 monotherapy arm in patients with AML or MDS and of the LGH447 + midostaurin treatment arm in patients with AML | weekly to bi-weekly up to 1.5 years
  Includes changes in hematology and blood chemistry values, assessments of physical examinations, vital signs, and electrocardiograms (ECGs)
PK parameters of the LGH447 monotherapy arm in patients with AML or MDS and of the LGH447 + midostaurin treatment arm in patients with AML | days 1, 2, 15, 16, 29, 30, 44, 57, and approximately monthly through Cycle 3
  LGH447 and midostaurin plasma concentrations and basic PK parameters
Changes between pre- and post-treatment levels of pS6RP and p4EBP1 in bone marrow aspirates and p4EBP1 in peripheral blood of the LGH447 monotherapy arm in patients with AML or MDS and of the LGH447 + midostaurin treatment arm in patients with AML | screening, days 1 and 29 up to 1.5 years
  Assess pharmacodynamic effects of LGH447
Anti-tumor activity in AML or high risk MDS associated wtih LGH447 | Day 29 up to 1.5 years
  To assess any preliminary anti-tumor activity in AML or high risk MDS associated with LGH447
Anti-tumor activity in AML or high risk MDS associated wtih LGH447 in combination with midostaurin | Day 29 up to 1.5 years
  To assess any preliminary anti-tumor activity in AML or high risk MDS associated with LGH447 in combination with midostaurin

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Novartis Investigative Site, Ann Arbor, Michigan, United States
- Novartis Investigative Site, Prahran, Victoria, Australia
- Novartis Investigative Site, Marseille, France
- Novartis Investigative Site, Ulm, Germany
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Shinagawa Ku, Tokyo, Japan
- Novartis Investigative Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLGH447X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17619